CLINICAL TRIAL: NCT05398289
Title: Four-week Duration Versus 6-week Duration of Therapy for the Treatment of Enterococcal Endocarditis
Brief Title: FOUR-SIX TRIAL for the Treatment of Enterococcal Endocarditis
Acronym: FOURSIX
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Alessandro Russo, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FST_2022
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Enterococcal Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4-week duration of antibiotic therapy (Experimental)
  Interventions: Drug: 4-week duration of antibiotic therapy
- standard 6-week duration of antibiotic therapy (Active Comparator)
  Interventions: Drug: 6-week duration of antibiotic therapy

INTERVENTIONS:
Drug: 4-week duration of antibiotic therapy — The aim is to show non-inferiority of a 4-week duration of antibiotic therapy versus a standard 6-week duration according to international guidelines
  Arms: 4-week duration of antibiotic therapy
Drug: 6-week duration of antibiotic therapy — The aim is to show non-inferiority of a 4-week duration of antibiotic therapy versus a standard 6-week duration according to international guidelines
  Arms: standard 6-week duration of antibiotic therapy

SUMMARY:
Duration of therapy in severe infections has a high impact in term of compliance, adverse events, and costs but also in term of antibiotic pressure on selection of multidrug-resistant pathogens. In this context, many advancements have been obtained for an early diagnosis of IE with a strict selection of criteria for surgery. Moreover, the use in antibiotic regimen of new drugs with peculiar PK/PD characteristics, as a quick bactericidal action, also for IE was not accompanied to a revaluation of duration of antibiotic treatment. On this basis, US and European guidelines recommend a 6-week duration of antibiotic treatment for IE due to enterococcal species.

AIM 1: To evaluate a 4-week duration of antibiotic therapy versus a 6-week duration according to international guidelines.

AIM 2: Second aim is to evaluate the PK/PD of antimicrobials in relation to the probability of target attainment (PTA) of optimal exposure against enterococci.

AIM 3: Finally, we will analyze the bactericidal activities of antibiotic combinations used in patients with IE and the survival of the subgroup of patients who underwent surgery.

Open-label, multicenter, randomized, non-inferiority trial to be conducted in a 3-year period. The institutional review board at each site will approve the protocol, and all patients or their authorized representatives will provide written informed consent. Eligible patients will be 18 years of age or older with a documented IE due to enterococcal strains, according to the modified Duke criteria.

63 patients in each of the two arms. The study will be conducted at Italian sites. Data on demographic characteristics, comorbidities, antibiotic and concomitant therapies will be collected. Baseline treatments will be defined according to the patients' pharmacological history. IE will be defined according to modified Duke criteria. Antibiotic treatment, indications and timing of surgery will be based on the 2015 American Heart Association and European Society of Cardiology guidelines.

Blood samples for determining antibiotic concentrations of ampicillin, gentamicin, vancomycin, daptomycin and linezolid will be collected at predetermined times in order to allow estimation of PK/PD.

Randomization:

1. 4-week duration of antibiotic therapy
2. standard 6-week duration of antibiotic therapy The intention-to-treat population (ITT) will include all randomized patients. The modified intention-to-treat population (mITT) will include all randomized patients receiving at least one dose of study medication. The clinically evaluable (CE) population will include ITT patients demonstrating sufficient adherence to study protocol.

Primary endpoint: non-inferiority of a 4-week course in terms of outcome at 60 days.

Secondary endpoints: microbiological eradication, pharmacological concentrations of antibiotic regimens, patients undergoing surgery, duration of therapy according with resistance profile of enterococcal species.

ELIGIBILITY:
Inclusion Criteria:

* documented infective endocarditis due to enterococcal strains, according to the modified Duke criteria.

Exclusion Criteria:

* patients candidate for chronic suppressive antibiotic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
A 4-week course of effective antimicrobial therapy | at 30 days and after 60 days from enrollment
  To evaluate clinical cure after 4 weeks of therapy

SECONDARY OUTCOMES:
Microbiological clearance of Enterococcus spp from blood cultures | From inclusion, up to 30 days
  Time to microbiological clearance from blood
Surgical Procedure | From inclusion, up to 30 days
  Time to surgery

IPD SHARING:
Plan to Share IPD: No